CLINICAL TRIAL: NCT02001727
Title: Long-term Effect of Screening and Eradication of Helicobacter Pylori in the General Population - HEP-FYN 12-years Follow-up
Brief Title: HEP-FYN 12-Years Follow-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Maria Bomme, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: s-20110054-97/262
Record Dates: First submitted 2013-09-16; First posted 2013-12-05 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Peptic Ulcer; Dyspepsia; Reflux
MeSH Terms: conditions — Peptic Ulcer; Dyspepsia; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hp-screened group (Active Comparator): Screened for Helicobacter Pylori and eradication therapy (1998-99)
  Interventions: Other: Questionaire
- Control group (Other): primarily unscreened group
  Interventions: Other: 13C-Urea breath test for Helicobacter Pylori; Other: Questionaire

INTERVENTIONS:
Other: 13C-Urea breath test for Helicobacter Pylori
  Arms: Control group
Other: Questionaire

SUMMARY:
Aims:

1. Evaluate the long-term effect of screening and eradication of Helicobacter Pylori on the prevalence of dyspepsia, and, as secondary outcomes, to assess the effect on dyspepsia related health-care consumption and quality of life.
2. To investigate symptoms of gastroesophageal reflux (GER), dyspepsia and the combination of these conditions and the effect on quality of life, prognosis and dyspepsia-related health care expenditure.

Methods:

In 1998-99 20.000 individuals, age 40-65 years, identified by their civil registration number, were allocated by a computerized randomized procedure to HP-screening group and control group. All participants received a questionnaire at inclusion, 1-year and 5-year and now again at 12 year follow-up assessing the prevalence of dyspepsia and quality of life. In addition we will obtain information from registers on, comorbidity, use of endoscopies and prescription medication. An economic evaluation is done alongside the randomized trial.

The primary unscreened group is invited to HP test (13C-urea breath-test) in order to analyze the effect of HP-screening according to HP-status

Expected results:

The study will provide information on the long-term effect of HP-screening and eradication in a population. The study will provide information about the long-term effect on incidence of peptic ulcer in an aging population that is likely to have an increased consumption of ASA and NSAID. Furthermore the study will generate knowledge about the long-term prognosis of dyspepsia and reflux in the population (dyspepsia and reflux. Preliminary results from the 5-yr follow-up (13) showed that is has a great influence on quality of life and the dyspepsia-related health care consumption, whether the individual has solely reflux, solely dyspepsia or a combination of both symptoms.

Long-term follow-up and further analyses of these findings could have great impact on management and treatment of individuals with symptoms. It is important to focus on groups; in which the symptoms have the greatest influence on quality of life of the individual. This finding has not been displayed in other studies.

DETAILED DESCRIPTION:
Questionnaire:

Information on abdominal symptoms (GRSR: Gastrointestinal symptom rating scale, rate of symptoms, quality of life (SF-36, EQ-5D-5L), consumption of ulcer drugs including over the counter drugs, hospital admissions, dyspepsia-related sick leave days, consultations and comorbidity). A reminder is sent out 2 weeks after the first contact.

Register data:

OPED (Odense Pharmaca-epidemiological Database): Information on reimbursable ulcer drugs, ASA, NSAID and HP-eradication therapy. The Regional Hospital discharge Register: Information based on International Classification of Diseases (ICD). Information on ulcer-related admissions, out-patient ulcer diagnosis and comorbidity, use of upper gastrointestinal endoscopy.

HP-test unscreened group:

Invitation of the primary unscreened group to HP test (13C-urea breath-test) in order to analyze the effect of HP-screening according to HP-status. Instruments: automated breath 13Co2 analyser- Isotope ratio mass spectrometer.

Almost all persons are infected with HP during childhood. Infection with the bacteria in adulthood is rare. Only few persons spontaneously turn HP-negative. From OPED we will know which individuals who have been prescribed HP-eradication treatment. Thus the participants in the control group, who are HP-positive at 12-yr follow-up, have had the infection the whole period. Provided they have not received HP-eradication treatment, those who are tested HP-negative have been so the whole period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals participating in 5 year follow-up

Exclusion Criteria:

* Individuals not participating in 5 year follow-up
* Moved outside the Region of Southern Denmark or with an unknown address
* Individuals who died

Ages: 52 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Economic Evaluation | twelve years
  The overall endpoint is expenditure in Danish kroner (on ulcer drugs, upper gastrointestinal endoscopy, GP consultations, hospital admissions related to peptic ulcer).
  Data on resource consumption of these services and procedures is multiplied with relevant unit prices, from the Danish Medicines Agency and the Danish National Board of Health, to assess a health-cost endpoint.

SECONDARY OUTCOMES:
Frequency of symptoms (dyspepsia, reflux) | twelve years
Drug consumption | Twelve years
  Consumption of ulcer drugs including over the counter drugs
Quality of life | twelve years
Incidence of esophagus- and gastric cancer | Twelve years
Upper gastrointestinal endoscopy / X-ray examinations of esophagus and gastric ventricle. | Twelve Years
Frequency of peptic ulcers incl. complicated ulcers | Twelve years

REFERENCES:
- [Derived] Bomme M, Hansen JM, Wildner-Christensen M, Hallas J, Schaffalitzky de Muckadell OB. Effects of Community Screening for Helicobacter pylori: 13-Year Follow-Up Evaluation of a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1715-1723.e7. doi: 10.1016/j.cgh.2017.06.006. Epub 2017 Jun 9. PMID 28606845